CLINICAL TRIAL: NCT02056327
Title: Phase One Study Evaluating Instrumentation for Dental Devices Used in Treating Sleep Apnea
Brief Title: Evaluating Instrumentation for Dental Devices Used in Treating Sleep Apnea
Status: Completed | Type: Observational
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Creare, Inc. (Industry)
Responsible Party: Principal Investigator, Glen P. Greenough, Assistant Professor of Neurology and Psychiatry, Dartmouth-Hitchcock Medical Center
Other Study IDs: HHSN268201300056C
Record Dates: First submitted 2014-02-04; First posted 2014-02-05 (Estimated); Last update posted 2014-03-27 (Estimated); Status verified 2014-03

CONDITIONS: Obstructive Sleep Apnea
Keywords: Oral Appliance
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Oral appliance with monitoring suite: Subjects will sleep with a standard oral appliance with the newly developed monitoring suite embedded within it for 1-2 nights while being monitored with standard in lab polysomnography or home sleep testing.
  Interventions: Device: A novel monitoring suite of sensors will be inserted into the standard oral device.

INTERVENTIONS:
Device: A novel monitoring suite of sensors will be inserted into the standard oral device.

SUMMARY:
Oral appliances are an accepted means to treat obstructive sleep apnea. We propose to develop monitoring sensors that could be inserted into commercially available oral appliances in order to monitor effectiveness of the oral appliances in treating sleep apnea.

DETAILED DESCRIPTION:
Oral appliances are an accepted means to treat obstructive sleep apnea. In order to determine if they are effective, a polysomnogram needs to be conducted with the oral appliance in place. We propose to develop monitoring sensors that could be inserted into commercially available oral appliances in order to monitor effectiveness of the oral appliances in treating sleep apnea. We propose to look at heart rate variability as a marker for ongoing sleep apnea. We will use temperature as means of detecting how long the device is in the mouth as a means of assessing adherence.

The objective of the Phase I project is to validate this hypothesis by answering five questions:

* What is the optimal sensor suite? We will determine the optimal suite of sensors that provides adequate sensitivity and specificity to determine OA usage and effectiveness without compromising patient comfort.
* Can we develop designs that are compatible with the most popular OAs? We will design and develop prototype versions of the OAMS that are compatible with three of the most popular commercially available OAMS products (potential candidates include EMA, TAP, SomnoDent, Herbst, Suad).
* Do experienced dental care providers who specialize in OAs approve of the designs? We will collaborate with dental care clinicians to iteratively refine the OAMS design for maximum performance and patient comfort.
* Does the OAMS provide data that are consistent with PSG instrumentation? We will collaborate with the Dartmouth-Hitchcock Medical Center (DHMC) Sleep Disorders Laboratory to assess OAMS sensor accuracy for approximately five healthy volunteers by comparing OSA-related OAMS data with data from standard PSG instrumentation.
* Can we formulate a cogent Human Subject Testing plan for Phase II? We will develop a detailed HST study plan to be conducted in Phase II to demonstrate fully integrated and functional OAMS in a broad range of OSA patients who are candidates for an OA.

ELIGIBILITY:
Inclusion Criteria:

* Ages 21-65
* Diagnosed with obstructive sleep apnea actively treated with an oral appliance or interested in transitioning to an oral appliance
* Ability to give informed consent

Exclusion Criteria:

* Significant physical illness that might impair the ability to participate
* Pregnant women will be excluded
* Subjects presently taking medication such as beta blockers or alpha agonists know to alter the autonomic nervous system

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults diagnosed with obstructive sleep apnea who are currently being treated with an oral appliance or who wish to transition to an oral appliance
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2013-11; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Polysomnography | One to two nights
  We will perform standard in-lab polysomnography or home sleep testing to assess the ability of the sensors embedded in the oral appliance to detect ongoing obstructive sleep apnea

CONTACTS AND LOCATIONS:
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States